CLINICAL TRIAL: NCT04102475
Title: Efficacy of a Phone-based Relapse Prevention for Anorexia Nervosa After a First Hospitalization
Acronym: EATLINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017_73; 2018-A02536-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eatline group (Experimental)
  Interventions: Other: Eatline
- control group (Sham Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Eatline — After discharge from a first hospitalization:
  Phone calls at 15 days, 1, 2, 4 and 9 months by a trained psychologist. The phone interview will be guided by the same standardized frame, which was developed by a group of experts and tested with a group of patients. The purpose of this intervention is to provide a therapeutic and motivational approach, with positive reinforcement and reassurance.
  * Added to treatment as usual (TAU): outpatient visits (at least monthly consultations) or scheduled hospitalizations
  * 6- and 12-month assessments as an outpatient interview with an assessor who is blind to condition
  Arms: eatline group
Other: Control — After discharge from the first hospitalization:
  * No specific phone calls
  * TAU: outpatient visits (at least monthly consultations) or scheduled hospitalizations
  * 6- and 12-month assessments as an outpatient interview with an assessor who is blind to condition
  Arms: control group

SUMMARY:
Anorexia Nervosa (AN) is a highly challenging disease which consequences are serious. Relapse rate is estimated between 38 and 41% during the year following hospitalization. The efficacy of patients' phone contact procedure on relapse has been assessed and has shown interest in numerous disorders. However, no study has ever used phone contact as a relapse prevention intervention tool in AN.

Objective: To evaluate efficacy of a phone contact procedure to increase body weight at 12 months after a first hospitalization for AN, by comparison to standard medical follow-up. Secondary objectives are to evaluate effect of phone contact procedure on: change in body weight at 6 month, general psychopathology disorder, psychopathology disorder specific to AN, rate of usual follow-up visit, and medico-economic impact.

Method: Prospective, multicenter, open-label, randomized controlled clinical trial, for subject over 15 years old presenting with diagnosis of AN. Patients randomized in EATLINE group will be contacted by phone at 15 days, 1, 2, 4 and 9 months after discharge from hospitalization. Patients in control group will benefit from usual follow-up.

Expected outcomes and perspectives:that there will be a significant decrease in relapse due to phone contact procedure compared to control group. Results would justify additional devices at the end of hospitalization, until development of various connected tools allowing to "stay in contact" with patients in order to optimize the current therapeutic possibilities of AN.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 15 years of age
* Diagnosis of AN (restrictive and/or purgative) according to DSM-5 criteria
* Included after a first inpatient hospitalization in specialized care
* Providing informed, dated and signed consent (for a minor, consent must be signed by both parents who have parental authority )
* With medical insurance
* Can be reached by telephone

Exclusion Criteria:

* Uncompensated psychiatric pathology
* Refusal to participate in the study
* The inability to consent to care (patient or his/her legal representative)
* Pregnancy
* Major incapable subject or under guardianship or judicial protection
* Homelessness
* No mastery of reading and writing

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
change in body mass index (BMI) | from discharge of the first hospitalization to 12 months.

SECONDARY OUTCOMES:
change in BMI from the first hospitalization | from the first hospitalization to 6 months and at 1 year
Mini International Neuropsychiatric Interview (MINI) | at baseline, at 6 months , at 1 year
SCID-2 (Structured Clinical Interview for DSM IV Axis II Personality Disorders) | at baseline, at 6 months , at 1 year
The level of psychopathology specific to AN assessed by EDI (Eating Disorders Inventory) | at baseline, at 6 months , at 1 year
The level of psychopathology specific to AN assessed BSQ (Body Shape Questionnaire) | at baseline, at 6 months , at 1 year
The level of psychopathology specific to AN assessed by WCS (Weight and Shape Concern Scale) | at baseline, at 6 months , at 1 year
Rate of patients lost to follow-up visits | during the one year
Rate of patients with at least one re-hospitalization or earlier consultations than expected | during the one year
Medico-economic evaluation with the MEDEC questionnaire | at 6 months, at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Cottencin, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (6):
- France (6):
  - Centre Hospitalier Général, Hénin-Beaumont
  - Hôpital Fontan2, CHU, Lille
  - Hôpital Saint Vincent de Paul, GHICL, Lille
  - Cliniqie Lautreamont, Loos
  - CHU de Montpellier, Montpellier
  - Centre Hospitalier Universitaire, Nantes